CLINICAL TRIAL: NCT06131970
Title: Effectiveness of Continuous Ketamine Infusion Associated With Magnesium Sulfate for Management of Patient With Chronic Pain : a Prospective Observational Study
Brief Title: The Effectiveness of Continuous Ketamine Infusion (KONTINUE)
Acronym: KONTINUE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Other Study IDs: 21-12
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain
Keywords: Pain; Neuropathic pain; Chronic pain; Fibromyalgia; Musculoskeletal diseases
MeSH Terms: conditions — Chronic Pain; Pain; Neuralgia; Fibromyalgia; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
There are different treatment for chronic pain. One possible treatment is intravenous infusions of ketamine.

DETAILED DESCRIPTION:
Ketamine continuous intravenous infusion for 4 days in Hospital with 0.5 mg/kg/day associated with Magnesium Sulfate 1000mg/day.

Evaluation schedules will be performed at day 15,30 and 60.

ELIGIBILITY:
Inclusion Criteria:

- Pain lasting for more than six months without contraindication to treatment

Exclusion Criteria:

* Inability to give consent
* Severe psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain treated with ketamine infusion
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Long-term effectiveness | 1 month
  Improvement of the numerical scale - score 0 to 10 - 10 is the worst
Long-term effectiveness | 1 month
  Clinical Global Impression of Change (CGI-C) - score 1 to 7 - 7 is the worst

SECONDARY OUTCOMES:
Pain relief | 15, 30, 60 days
  Neuropathic Pain Symptom Inventory (NPSI) - score 0 to 10 - 10 is the worst
Variation of quality of life | 15, 30, 60 days
  Short Form 12 health survey
Variation of quality of life | 15, 30, 60 days
  Hospital Anxiety and Depression scale - score 0 to 21 - 21 is the worst

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No